CLINICAL TRIAL: NCT04670159
Title: The Effectiveness of Online Physical Activity and Ergonomics Training in Physiotherapy Students Receiving Distance Education
Brief Title: Online Physical Activity and Ergonomics Training in Physiotherapy Students Receiving Distance Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilay Arman, Assistant Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10832
Record Dates: First submitted 2020-12-06; First posted 2020-12-17 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Health Behavior; Ergonomics; Online Education
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Education Group (Experimental)
  Interventions: Behavioral: Online Education
- Brochure Group (Experimental)
  Interventions: Behavioral: Information With Brochure

INTERVENTIONS:
Behavioral: Online Education — Online ergonomics, exercise and physical activity training will be provided 3 times a week for 6 weeks. The trainings it is planned to be made with a video-based online platform called Edpuzzle. With the online classroom created, the student education will be provided. A total of 18 training videos will be prepared, each video is 6-10 minutes. After the training there will be an individual motivational interview with the students in the this group with the zoom application. With motivational interview solutions by revealing the willingness, obstacles and indecision of the student to transfer the learned information to his daily life will be recommended.
  Arms: Online Education Group
Behavioral: Information With Brochure — An e-brochure will be prepared for students in this group to provide information on ergonomics, physical activity and exercise. and the e-brochure will be sent to the students via e-mail after the initial evaluation.
  Arms: Brochure Group

SUMMARY:
The pandemic process has caused very important changes and effects in the economy, social life and education practices, especially health at global level. Within the scope of the measures taken, with the closure of educational institutions and interruption of face-to-face education, the education of 1.6 billion students, which corresponds to approximately half of the student population from all educational levels, has been interrupted. The need and approach to open and distance learning has come to the fore with significant changes and effects on education worldwide. Pandemic measures, the transition to distance education and the increase in computer usage caused an increase in ergonomic risks in students. Due to the pandemic process, it has been reported that the physical activity level of students decreases and the sitting period is prolonged. In this study, physiotherapy students who receive distance education will be given online ergonomics and physical activity training and the results will be evaluated.

DETAILED DESCRIPTION:
The pandemic process has caused very important changes and effects in the economy, social life and education practices, especially health at global level. Within the scope of the measures taken, with the closure of educational institutions and interruption of face-to-face education, the education of 1.6 billion students, which corresponds to approximately half of the student population from all educational levels, has been interrupted. The need and approach to open and distance learning has come to the fore with significant changes and effects on education worldwide. Pandemic measures, the transition to distance education and the increase in computer usage caused an increase in ergonomic risks in students. Due to the pandemic process, it has been reported that the physical activity level of students decreases and the sitting period is prolonged. In this study, physiotherapy students who receive distance education will be given online ergonomics and physical activity training and the results will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being receiving distance education due to the Covid pandemic
* Being in the age range of 18-25

Exclusion Criteria:

* Congenital or subsequent disability affecting the musculoskeletal system
* Presence of cognitive impairment
* Having a diagnosed psychiatric disorder
* Having a neurological or cardiovascular disease
* Exercising regularly

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-12-06 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Change in ergonomic risks in the distance education process | Baseline, change from baseline ergonomics risks levels at 6 weeks
  The ergonomic risk levels of the participants in the distance education process will be determined by Rapid Office Strain Assessment (ROSA) .The Rapid Office Strain Assessment (ROSA) was designed to quickly quantify risks associated with computer work and to establish an action level for change based on reports of worker discomfort. Ergonomic risk assessment will be done after online training and brochure information for all participants.

SECONDARY OUTCOMES:
Measuring the prevalence of musculoskeletal disorder By Cornell questionniare Questionnaire | Baseline, 6 weeks
  The Cornell Musculoskeletal Discomfort Questionnaire is an outcome measure used widely when examining musculoskeletal disorders in various occupational groups and students alike.The Cornell Musculoskeletal Discomfort Questionnaire was taken from the instruments provided by Human Factors and Ergonomics Laboratory at Cornell University.
  The changes in the musculoskeletal disorders of the participants will be evaluated before and after the online training and brochure information.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpaşa, Istanbul, Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No